CLINICAL TRIAL: NCT04863547
Title: Severity of the New UK SARS-Cov2 Variant in COVID-19 Infection
Acronym: SEVASAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 0007S SEVASAR
Record Dates: First submitted 2021-04-08; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Patients hospitalized for COVID-19 with SARS-CoV-2 variant 20I / 501Y.V1
  Interventions: Other: Data collection
- Non exposed: Patients hospitalized for COVID-19 to SARS-CoV-2 corresponding to wild type 20A variants. EU1 or 20A. EU2
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
The COVID-19 epidemic has now raged for more than a year with more than 100 million identified cases and nearly 2.5 million deaths worldwide. Since November 2020, we have been witnessing the emergence of viral variants in different regions of the world. This expected genetic drift of the virus, but somewhat abrupt since November, raises questions concerning the characteristics of transmissibility, pathogenicity, sensitivity to possible treatments, and escape from natural or vaccine immunity. The objective of this study is to find out whether the new variants of SARS-CoV-2 are associated with particular clinical forms. The results of this research will provide elements to determine whether the new variants of SARS-CoV-2 are associated with more severe clinical forms.

DETAILED DESCRIPTION:
SEVASAR is a paired cohort study with retrospective data collection:

* Presentation: patients hospitalized for COVID-19 with SARS-CoV-2 variant 20I / 501Y.V1
* Not exposed: patients hospitalized for COVID-19 with SARS-CoV-2 corresponding to wild variants type 20A. EU1 or 20A. EU2

The severity of illness will be compared between pairs. Disease severity will be assessed according to the following definition: defined by a composite criterion including, at 28 days after hospital admission: WHO scale >5 /11 levels, (death OR need for invasive ventilation OR need for high flow ventilation (Optiflex or NIV or CPAP) or high concentration mask. This event will be taken into account regardless of its time of occurrence between the first day of the hospitalization studied and D29 after hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Acute symptomatic PCR + COVID with screening
* Hospitalized for acute COVID between 01/01/2021 (or since the setting up of the screening in the center) and 02/28/2021

Exclusion Criteria:

* Opposition to participation
* Identification of variants other than 20I / 501Y.V1
* Patients infected with SARS-CoV-2 in a nosocomial context

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Acute symptomatic COVID PCR+ with screening Hospitalized for acute COVID between January 1,2021 (or since the implementation of the screening in the center) and february 28, 2021
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
To estimate the proportion of Severe disease form | between the first day of hospitalization and Day 29
  Percentage of severe form. Severity was defined by a composite criterion including, at Day 28 days from hospital admission: WHO scale >5 /11 levels, (death OR required invasive ventilation OR required high flow ventilation (Optiflex or NIV or CPAP) or high concentration mask.
To estimate the proportion of Mortality | Day 29
  Percentage of mortality
To estimate the proportion of WHO score > 5 | between the first day of hospitalization and Day 29
  Percentage of WHO score > 5
To estimate the proportion of Patient who received critical care | between the first day of hospitalization and Day 29
  Percentage of patients who received critical care
To estimate the proportion of patients who had invasive ventilation | between the first day of hospitalization and Day 29
  Percentage of patients who had invasive ventilation
To estimate the proportion of patients who had high flow oxygen therapy | between the first day of hospitalization and Day 29
  Percentage of patients who had high flow oxygen therapy
Time between the first day of symptoms and the first day of hospitalization | between first day of symptoms and the first day of hospitalization assessed up to one month
  Time between the first day of symptoms and the first day of hospitalization
Delay between the first day of symptoms and the first day of hospitalization | between first day of symptoms and the first day of hospitalization assessed up to one month
  Time between the first day of symptoms and the first day of hospitalization
Time between the first day of symptoms and the severity of disease | between first day of symptoms and the severity assessed up to one month
  Time between the first day of symptoms and the severity of disease
Time between the first day of symptoms and mortality | between first day of symptoms and mortality assessed up to two month
  Time between the first day of symptoms and mortality

CONTACTS AND LOCATIONS:
Locations (53):
- France (52):
  - CHU Amiens Picardie Site Nord, Amiens
  - CHU Angers, Angers
  - Centre hospitalier de Béziers, Béziers
  - hôpital Avicenne, Bobigny
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Centre hospitalier métropole Savoie, Chambéry
  - Centre Hospitalier Châteaubriant Nozay Pouancé, Châteaubriant
  - Hôpital Beaujon, Clichy
  - Hôpitaux Civils de Colmar, Colmar
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Centre hopsitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Intercommunal, Créteil
  - Hôpital Henry Mondor, Créteil
  - CHU Dijon Bourgogne, Dijon
  - Hôpital de Garches, Garches
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital SALENGRO, Lille
  - CHU Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier François Quesnay, Mantes-la-Jolie
  - Hôpital André Grégoire, Montreuil
  - Hopital Confluent, Nantes
  - CHU Nantes, Nantes
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hôpital Archet, Nice
  - Hôpital Carémeau, Nîmes
  - Centre Hospitalier du Centre-Bretagne, Noyal-Pontivy
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - HôpitalSaint Antoine, Paris
  - hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Hôpital Bichat, Paris
  - Hôpital Tenon, Paris
  - Hôpital Saint Louis, Paris
  - Centre hospitalier de Perigueux, Périgueux
  - CHI de Poissy/Saint-Germain-en-Laye, Poissy
  - CHU, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicoll, Rouen
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - Nouvel Hopital Civil, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital Purpan, Toulouse
  - Centre hospitalier de Tourcoing, Tourcoing
  - CHU Tours, Tours
  - Centre Hospitalier de Valence, Valence
  - Centre hospitalier de Valenciennes, Valenciennes
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Institut Gustave Roussy, Villejuif
  - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges
- André Zobda Cabié, Fort-de-France, Martinique France, Martinique

IPD SHARING:
Plan to Share IPD: Undecided